CLINICAL TRIAL: NCT05145608
Title: Single Dose Two Way Crossover Comparative Bioavailability Study of Lamotrigine Extended-Release Tablets USP 50 mg in Healthy Male and Female Volunteers Fasting State
Brief Title: Comparative Bioavailability Study of Lamotrigine ER Tablets USP 50 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alembic Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AMC-P0-215
Record Dates: First submitted 2018-01-09; First posted 2021-12-06 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Intervention Model Description: Single center, randomized, single dose, laboratory-blinded, 2-period, 2-sequence, crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test- Lamotrigine ER Tablets USP 50mg (Active Comparator): Single dose of Test- Lamotrigine ER Tablets USP 50mg will be administered
  Interventions: Drug: Lamotrigine ER tablet 50mg
- Reference- Lamictal® XRTM ER tablet 50mg (Active Comparator): Single dose of Reference- Lamictal® XRTM (Lamotrigine) ER tablet 50mg will be administered
  Interventions: Drug: Lamotrigine ER tablet 50mg

INTERVENTIONS:
Drug: Lamotrigine ER tablet 50mg — In each study period, a single 50 mg dose of lamotrigine will be administered orally with about 240 mL of water at ambient temperature, in the morning, while subjects are seated, following a 10-hour overnight fast.
  Other Names: Reference- Lamictal® XRTM (Lamotrigine) ER tablet 50mg

SUMMARY:
Objective:

To evaluate and compare the bioavailability and therefore to assess the bioequivalence of two different formulations of lamotrigine after a single oral dose administration under fasting conditions.

The secondary objective is to monitor the safety of the subjects.

DETAILED DESCRIPTION:
Study Design:

Single center, randomized, single dose, laboratory-blinded, 2-period, 2-sequence, crossover design

Subjects:

Twenty-two (22) subjects will be included in the study.

Main Inclusion Criteria:

Male and female volunteers, non- or ex-smokers, of at least 18 years of age to 54 years of age, inclusively, with a body mass index (BMI) within 22.00 to 30.00 kg/m2, inclusively, with a minimum body weight of 60 kg, will be selected according to the inclusion and exclusion criteria.

Blood Sampling:

In each study period, 23 blood samples will be collected. The first blood sample will be collected prior to drug administration while the others will be collected up to 192 hours after the drug administration.

Wash-out:

The drug administrations will be separated by at least 28 calendar days.

Tests during study:

An alcohol breath test will be performed before each period of the study. Screening for drugs of abuse will be performed before each period of the study. A C-SSRS questionnaire will be performed prior to each study period, as well as prior to discharge for each period of the study.

For female subjects, a serum pregnancy test will be performed before each period of the study.

Vital signs will be measured prior to and approximately 2, 4, 8, 10, 12, 24, 36 and 48 hours following each drug administration.

Neurological function tests will be performed approximately 30 hours after each drug administration.

For safety reasons, hematology tests will be performed before the 2nd period of the study.

Post study Tests:

Hematology, general biochemistry (including a serum pregnancy test for female subjects), and urinalysis tests will be repeated along with the collection of the last blood sample of the study.

A complete physical examination (including vital signs) will also be performed.

Bioanalysis: Lamotrigine plasma concentrations will be measured by a validated bioanalytical method.

ELIGIBILITY:
Inclusion Criteria:

1. Availability for the entire study period
2. Motivated volunteer and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the physician or designee
3. Male or female volunteer
4. A female volunteer must meet one of the following criteria:

   1. Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first administration of the study drug, during the study and for at least 30 days after the last dose of the study drug. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Intrauterine device (without hormones)
      * Condom with intra-vaginally applied spermicide or
   2. Participant is of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses)
5. Volunteer aged of at least 18 years to 54 years of age, inclusively
6. Volunteer with a BMI within 22.00 to 30.00 kg/m2, inclusively
7. Minimum body weight of 60 kg
8. Non- or ex-smokers; an ex-smoker being defined as someone who completely stopped smoking for at least 6 months before day 1 of this study
9. Clinical laboratory values within the laboratory's stated normal range; if not within this range, must be without any clinical significance
10. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, general biochemistry, ECG and urinalysis)
11. Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer The informed consent form must be signed by all volunteers prior to their participation in the study.

Exclusion Criteria:

1. Difficulty donating blood
2. History of difficulty in swallowing or of any gastrointestinal disease which could affect drug absorption
3. Volunteer who is associated to Algorithme Pharma (staff member or immediate family of a staff member)
4. Females who are pregnant or are lactating
5. History of significant hypersensitivity to lamotrigine or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
6. History of any prior allergic drug rash
7. Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
8. History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
9. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
10. Showing suicidal tendency as per the Columbia Suicide Severity Rating Scale (C-SSRS) administered at screening
11. Presence of out-of-range cardiac interval (PR < 110 msec, PR > 220 msec, QRS < 60 msec, QRS >119 msec and QTc > 450 msec for males and > 460 msec for females) on the screening ECG or other clinically significant ECG abnormalities
12. Known presence of rare hereditary problems of galactose and /or lactose intolerance, lactase deficiency or glucose-galactose malabsorption
13. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
14. Any clinically significant illness in the previous 28 days before day 1 of this study
15. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin and St John's Wort), in the previous 28 days before day 1 of this study
16. Any history of tuberculosis and/or prophylaxis for tuberculosis
17. Positive screening of alcohol and/or drugs of abuse
18. Positive results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or Hepatitis C Virus (HCV (C)) tests
19. Females who are pregnant according to a positive serum pregnancy test
20. Volunteers who took an Investigational Product (in another clinical trial) in the previous 28 days before day 1 of this study
21. Volunteers who took an Investigational Product (in another clinical trial) with a long half-life (≥120 hours) in the previous 3 months before day 1 of this study
22. Volunteers who took lamotrigine in the previous 28 days before day 1 of this study
23. Females who use the following systemic contraceptives: oral, patch or vaginal ring, in the 28 days before day 1 of this study
24. Females who use hormone replacement therapy in the 28 days before day 1 of this study
25. Females who use the following systemic contraceptives: injections or implant, or hormone-releasing intrauterine device in the previous 13 weeks before day 1 of this study
26. Volunteers who donated 50 mL or more of blood in the previous 28 days before day 1 of this study
27. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 192 hours
  Peak Plasma Concentration (Cmax)
AUC0-T | Up to 192 hours
  Area under the plasma concentration versus time curve (AUC)
AUC0-∞ | Up to 192 hours
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma, Mount Royal, Quebec, Canada